CLINICAL TRIAL: NCT06054672
Title: Effect of Subthreshold Stimulation on Pain and Muscle Activity in Patients With Chronic Low Neck Pain and Myofascial Trigger Points
Brief Title: Subthreshold Stimulation on Chronic Low Neck Pain Myofascial Trigger Points
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Ayman Mohamed, Assistant Lecturer, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Beni-Suef University 1
Record Dates: First submitted 2023-09-08; First posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Chronic Neck Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): This group will receive subthreshold stimulation
  Interventions: Device: Subthreshold Electrical stimulation
- Group II (No Intervention): This group will receive no stimulation

INTERVENTIONS:
Device: Subthreshold Electrical stimulation — We will use a electrotherapy device to deliver subthreshold Electrical stimulation
  Arms: Group 1

SUMMARY:
This study will investigate the effect of subthreshold stimulation on pain and muscle activity in patients with chronic low neck pain and myofascial trigger points.

DETAILED DESCRIPTION:
The study will include 2 groups. One group will receive subthreshold stimulation and other will not receive any treatment. The measurements will include pain and myscle activity.

ELIGIBILITY:
Inclusion Criteria:

* chronic neck pain
* One or more trigger point

Exclusion Criteria:

* any musculoskeletal or neuromuscular diseases

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2023-09-30 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Electromyographical signals | 2 months
  We will record the the Trapezius muscle activity of both sides.
Pressure sensitivity using pressure ergometer | 2 months
  We will measure pain threshold produced from Trapezius muscle

SECONDARY OUTCOMES:
Neck pain and disability | 2 months
  We will record the level of pain and disability in neck using neck pain and disability index. standard instrument for measuring self-rated disability due to neck pain and is used by both clinicians and researchers. Each of the 10 items scores from 0 to 5. The maximum score is 50. The obtained score can be multiplied by two to produce a percentage score
Functional ability | 2 months
  We will measure the functional ability. The Copenhagen Neck Functional Disability Scale has been developed for those who have neck pain and disabilities due to the pain. The scale includes questions relating to headache, ability to sleep and to concentrate and activities of daily living.